CLINICAL TRIAL: NCT03783546
Title: Acupuncture for Hot Flashes in Hormone Receptor-Positive Breast Cancer, a Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: The Comprehensive and Integrative Medicine Institute of South Korea (Other)
Responsible Party: Principal Investigator, Weidong Lu, MB, MPH, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-371
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Immediate Acupuncture (Experimental): * Will receive a standardized acupuncture protocol for a 10-week period
  * 20 sessions: twice a week for 10 weeks
  * After the completion of the 10 weeks main study period, participants will cross over to the usual care as a follow-up without acupuncture for additional 10 weeks.
  Interventions: Device: Acupuncture
- Delayed acupuncture (Active Comparator): * Will receive standard usual care without acupuncture for 10 weeks
  * Participants will cross over to receive the same acupuncture protocol for 10 weeks --10 sessions: once a week for 10 weeks before exiting the study
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Acupuncture — Acupuncture is a complementary therapy in which, hair-thin, sterile disposable needles are inserted into various spots on your skin, with the goal of affecting body's natural healing system
  Arms: Immediate Acupuncture
Other: Usual Care — the current standard of care with non-hormonal pharmacotherapy of western medicine
  Arms: Delayed acupuncture

SUMMARY:
This research study is evaluating acupuncture, a medical therapy in which hair-thin, stainless steel needles are shallowly inserted into specific points to help the body's natural healing process, as a possible treatment to reduce hot flashes.

DETAILED DESCRIPTION:
Hot flashes are a sensation of sudden onset of body warmth, flushing and sweating. Hot flashes are common side effects of breast cancer treatments and can affect mood and daily life. Medications can help ease hot flashes, but many patients continue to experience symptoms despite these treatments.

Acupuncture is a complementary therapy in which, hair-thin, sterile disposable needles are inserted into various spots on the skin, with the goal of affecting body's natural healing system. Acupuncture has been tested in clinical trials in cancer patients and has been shown to be helpful in treating a number of side effects of cancer treatment, such as nausea and vomiting from chemotherapy. A few early studies have suggested that acupuncture may help to lessen hot flashes, but more information is needed about the benefits of acupuncture in breast cancer patients.

This study is being done to test whether acupuncture can help to reduce the number and intensity of hot flashes in breast cancer patients who are being treated with mediations such as tamoxifen and aromatase inhibitors, such as anastrozole (Arimidex), exemestane (Aromasin), and letrozole (Femara).

ELIGIBILITY:
Inclusion Criteria:

* History of histologically or cytologically proven Stage I-III breast cancer with estrogen receptor positive with HER-2 positive or negative tumor;
* Premenopausal or postmenopausal status;
* Completed all primary chemotherapy and surgery;
* Currently undergoing adjuvant hormonal therapy (e.g. Tamoxifen and/or Aromatase inhibitors) with or without ovarian function suppression for at least 4 weeks at study entry; the use of Trastuzumab after adjuvant chemotherapy is allowed;
* Reported persistent hot flashes for at least 4 weeks AND more than 14 episodes of hot flashes per week (2 hot flashes per day) during the week prior to the study entry;
* Age ≥ 18 years;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Signed informed consent

Exclusion Criteria:

Undergoing chemotherapy or planned surgery, chemotherapy, change doses and regimen of hormonal therapy during the study period;

* Unstable cardiac disease or myocardial infarction within 6 months prior to study entry;
* Uncontrolled seizure disorder or history of seizure;
* Active clinically significant uncontrolled infection;
* Use of acupuncture for hot flashes within 6 months prior to the study entry;
* Uncontrolled major psychiatric disorders, such as major depression or psychosis;
* Newly starting pharmacologic treatment of hot flashes such as selective serotonin reuptake inhibitors (SSRIs) and/or anti-convulsant for less than 4 weeks prior to study entry. Participants may continue with medications or therapies for the treatment of hot-flashes while participating in the study if the medication has been taking for more than 4 weeks prior to study entry AND the dose of the medication is going to be kept consistently during the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2025-12-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Lu, PhD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor- Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Requests may be directed to: [contact information for Sponsor- Investigator or designee].

REFERENCES:
- [Derived] Baedorf Kassis S, Lu W, White SA, Shin IH, Park SH, Jeong YJ, Yao C, Ligibel J, Bierer BE. Developing and implementing a self-monitoring toolkit for a coordinated multinational randomized acupuncture trial. BMC Complement Med Ther. 2022 Jun 17;22(1):161. doi: 10.1186/s12906-022-03648-4. PMID 35715806

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 84 patients consented, and 78 patients were randomized.
Pre-assignment Details: Enrollment: Accrual began in January-February 2019. DFCI site suspended study accrual for several months during the COVID-19 pandemic and resumed when approved by local authorities. DFCI completed accrual in June 2021, meeting its accrual goal. Due to the pandemic, 84 patients who consented to participate but 6 were not able to be randomized to the study therapy.
Groups:
- Immediate Acupuncture: * received a standardized acupuncture protocol for a 10-week period
  * 20 sessions: twice a week for 10 weeks
  * After the completion of the 10 weeks main study period, participants crossed over to the usual care as a follow-up without acupuncture for additional 10 weeks.
  Acupuncture: Acupuncture is a complementary therapy in which, hair-thin, sterile disposable needles are inserted into various spots on your skin, with the goal of affecting body's natural healing system
- Delayed Acupuncture: * received standard usual care without acupuncture for 10 weeks
  * Participants crossed over to receive the same acupuncture protocol for 10 weeks --10 sessions: once a week for 10 weeks before exiting the study
  Usual Care: the current standard of care with non-hormonal pharmacotherapy of western medicine
Period: Overall Study
Arm/Group | Immediate Acupuncture | Delayed Acupuncture
Started | 39 | 39
Completed | 35 | 36
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Delayed Acupuncture: * received standard, usual care without acupuncture for 10 weeks
  * Participants crossed over to receive the same acupuncture protocol for 10 weeks --10 sessions: once a week for 10 weeks before exiting the study
  Usual Care: the current standard of care with non-hormonal pharmacotherapy of western medicine
- Total: Total of all reporting groups
Arm/Group | Immediate Acupuncture | Delayed Acupuncture | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.3 (11.2) | 47.7 (7.7) | 49 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 39 | 78
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 33 | 30 | 63
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 39 | 78
Hot Flash Score [Mean (Standard Deviation); unit: HFS units on a scale] — It is a validated and reliable method for collecting subjective data on both the frequency and severity of hot flashes. Participants are asked to record the frequency and severity of hot flashes each day on a scale ranging from 1 to 4 (1 = mild, 2 = moderate, 3 = severe, 4 = very severe). The mean Hot Flash Score (HFS) is calculated by multiplying the frequency by the severity of hot flashes recorded in the daily diary.
  HFS units on a scale | 9.5 (6.8) | 11.0 (7.2) | 10.25 (7.0)
ESS of FACT-ES [Mean (Standard Deviation); unit: units on a scale] — The Endocrine Symptom Subscale (ESS) of the Functional Assessment of Cancer Therapy-Endocrine Symptoms (FACT-ES) is validated scale that contains 19 items that specifically assess endocrine symptoms, including hot flashes, night sweats, vaginal dryness, and joint pain, with scores ranging from 0-76. Lower scores indicate worse endocrine symptoms.
  units on a scale | 50.0 (8.8) | 51.6 (8.5) | 50.8 (8.65)
FACT-B Total Score [Mean (Standard Deviation); unit: FACT-B total score] — The Functional Assessment of Cancer Therapy - Breast (FACT-B) is a 37-item instrument designed to measure five domains of quality of life in breast cancer patients: Physical (PWB), social (SWB), emotional (EWB), functional well-being (FWB), as well as a breast-cancer subscale (BCS). The response values for each question range from 0 (not at all) to 4 (very much). Higher scores on any subscale suggest better quality of life. Final scores (FACT-B-Total) of all subscales range from 0 to 148, where 148 represents the most favorable score and the highest QoL.
  FACT-B total score | 102.5 (17.9) | 103.6 (16.3) | 103.05 (17.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Weekly HFS Score Between Acupuncture and Usual Care Arms at the End of Week 10
Description: Daily Hot Flash Diary (DHFD) The DHFD is a measure of self-reported hot flash data that uses a diary to record the frequency and severity of hot flashes based on a 4-point scale (i.e., mild, moderate, severe, or very severe) to provide a hot flash score/index that reflects both number and severity of hot flashes (i.e., sum of the number of hot flashes multiplied by a weighted severity). Patients were asked to record daily for a week at five time points through the trial: baseline, week 5, week 10, week 15, and week 20. Negative changes would suggest improvements in number, type, or severity.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: HFS score on a scale
Groups:
- Immediate Acupuncture: * received a standardized acupuncture protocol for a 10-week period
  * 20 sessions: twice a week for 10 weeks
  * After the completion of the 10-week main study period, participants crossed over to the usual care as a follow-up without acupuncture for additional 10 weeks.
  Acupuncture: Acupuncture is a complementary therapy in which, hair-thin, sterile disposable needles are inserted into various spots on your skin, with the goal of affecting body's natural healing system
Arm/Group | Immediate Acupuncture | Delayed Acupuncture
Number analyzed (Participants) | 29 | 30
HFS score on a scale | -5.3 (3.9) | -0.5 (6.5)
Statistical Analysis 1: Comparison: Immediate Acupuncture vs Delayed Acupuncture; Test type: Superiority; p = 0.0003, Mixed Models Analysis

2. Secondary Outcome: Changes in the Total and Subscores in Functional Assessment of Cancer Therapy- Breast Cancer
Description: Changes in scores were calculated as (Week-10 - baseline). Since a higher score on any FACT-B subscale indicates better quality of life, a positive change would suggest that the patient's score improved during that time interval.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: FACT-B total score
Arm/Group | Immediate Acupuncture | Delayed Acupuncture
Number analyzed (Participants) | 29 | 30
FACT-B total score | 6.6 (11.3) | -1.9 (8.4)

3. Secondary Outcome: Changes in the Endocrine Symptom Subscale (ESS) in Functional Assessment of Cancer Therapy- Endocrine Symptoms (FACT-ES)
Description: The ESS is one subscale of the FACT-ES that assesses hormonal symptoms of endocrine therapy. The score ranges from 0-76 with higher scores indicating greater freedom from symptoms. Changes in scores were calculated as (Week-10 - baseline). Since a higher score reflects increased freedom from hormonal symptoms, a positive change would suggest that the patient's symptoms improved during that time interval.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: ESS score on FACT-ES
Groups:
- Immediate Acupuncture: * Will receive a standardized acupuncture protocol for a 10-week period
  * 20 sessions: twice a week for 10 weeks
  * After the completion of the 10 weeks main study period, participants will cross over to the usual care as a follow-up without acupuncture for additional 10 weeks.
  Acupuncture: Acupuncture is a complementary therapy in which, hair-thin, sterile disposable needles are inserted into various spots on your skin, with the goal of affecting body's natural healing system
- Delayed Acupuncture: * Will receive standard usual care without acupuncture for 10 weeks
  * Participants will cross over to receive the same acupuncture protocol for 10 weeks --10 sessions: once a week for 10 weeks before exiting the study
  Usual Care: the current standard of care with non-hormonal pharmacotherapy of western medicine
Arm/Group | Immediate Acupuncture | Delayed Acupuncture
Number analyzed (Participants) | 29 | 30
ESS score on FACT-ES | 5.3 (7.0) | -0.5 (6.6)
Statistical Analysis 1: Comparison: Immediate Acupuncture vs Delayed Acupuncture; Test type: Superiority; p = 0.002, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 20 weeks: The adverse events were reported separately for each intervention phase to accurately capture the effects of the treatments. The study had two arms: Immediate Acupuncture Arm (Treatment Weeks 1-10) and (Usual Care Weeks 11-20) Adverse events were recorded during both the treatment and follow-up phases. Delayed Acupuncture Arm (Usual Care Weeks 1-10) and (Intervention Weeks 11-20) Adverse events were recorded during both the usual care and intervention phases.
Groups:
- Immediate Acupuncture (Treatment Weeks 1-10): * received a standardized acupuncture protocol for a 10-week period
  * 20 sessions: twice a week for 10 weeks
  * After the completion of the 10 weeks main study period, participants crossed over to the usual care as a follow-up without acupuncture for additional 10 weeks.
  Acupuncture: Acupuncture is a complementary therapy in which, hair-thin, sterile disposable needles are inserted into various spots on your skin, with the goal of affecting body's natural healing system
- Delayed Acupuncture (Usual Care Weeks 1-10): * received standard usual care without acupuncture for 10 weeks
  * Participants crossed over to receive the same acupuncture protocol for 10 weeks --10 sessions: once a week for 10 weeks before exiting the study
  Usual Care: the current standard of care with non-hormonal pharmacotherapy of western medicine
- Immediate Acupuncture (Usual Care Weeks 11-20): -After the completion of the 10 weeks main study period, participants crossed over to the usual care as a follow-up without acupuncture for additional 10 weeks.
- Delayed Acupuncture (Intervention Weeks 11-20): -Participants crossed over to receive the same acupuncture protocol for 10 weeks
  --10 sessions: once a week for 10 weeks before exiting the study
Arm/Group | Immediate Acupuncture (Treatment Weeks 1-10) | Delayed Acupuncture (Usual Care Weeks 1-10) | Immediate Acupuncture (Usual Care Weeks 11-20) | Delayed Acupuncture (Intervention Weeks 11-20)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39 | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 2/39 | 0/39 | 0/39 | 0/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Acupuncture (Treatment Weeks 1-10) (N=39) | Delayed Acupuncture (Usual Care Weeks 1-10) (N=39) | Immediate Acupuncture (Usual Care Weeks 11-20) (N=39) | Delayed Acupuncture (Intervention Weeks 11-20) (N=39)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — 1 case grade-2 pain; 1 case grade-1 heart palpitations
heart palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — grade-1 heart palpitations

LIMITATIONS AND CAVEATS:
We randomized patients to immediate acupuncture vs. delayed acupuncture rather than using an active control condition. This raises the possibility that the placebo effect could have contributed to the impact of the immediate acupuncture intervention on hot flashes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-03): https://cdn.clinicaltrials.gov/large-docs/46/NCT03783546/Prot_SAP_000.pdf